CLINICAL TRIAL: NCT01945840
Title: Do Gut Hormones Mediate the Beneficial Effects of Roux-en-Y Bypass?
Brief Title: Gut Hormones and Roux en Y Gastric Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MR/K02115X/1
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Roux en Y Gastric Bypass (Active Comparator): Participants will be those already scheduled to undergo Roux en Y Gastric Bypass Surgery
  Interventions: Procedure: Roux en Y Gastric Bypass Surgery
- Gut hormone infusion (Experimental): Infusion of three gut hormones (GLP-1, PYY and oxyntomodulin) subcutaneously for 4 weeks as below:
  * Combination of GLP-1/OXM/PYY (GOP)
  * Single GLP-1
  * Single OXM
  * Single PYY
  * Combination of GLP-1 and OXM
  * Combination of GLP-1 and PYY
  * Combination of OXM and PYY
  Interventions: Other: Gut hormone infusion
- Placebo infusion (Placebo Comparator): Saline infusion given subcutaneously for 4 weeks.
  Interventions: Other: Placebo infusion
- Very low calorie diet (Active Comparator): Participants will be asked to follow a very low calorie diet for 4 weeks.
  Interventions: Other: Very low calorie diet

INTERVENTIONS:
Procedure: Roux en Y Gastric Bypass Surgery
  Arms: Roux en Y Gastric Bypass
Other: Gut hormone infusion
  Arms: Gut hormone infusion
Other: Placebo infusion
  Arms: Placebo infusion
Other: Very low calorie diet
  Arms: Very low calorie diet

SUMMARY:
The purpose of this study is to assess whether the changes in gut hormones seen following Roux en Y Gastric Bypass surgery are responsible for some of the beneficial effects seen post-operatively.

DETAILED DESCRIPTION:
This study is designed to investigate whether chronic elevation of glucagon-like peptide-1 (GLP-1), oxyntomodulin and peptide YY (PYY) in combination is responsible for the majority of the metabolic effects of Roux-en-Y gastric bypass (RYGB) including improved glycaemia, increased energy expenditure, reduced food intake, weight loss, reduced preference for high calorie foods and reduced activation in brain reward areas in response to visual food cues.

ELIGIBILITY:
Inclusion criteria

* Aged 18 - 70 years.
* Male or female.
* Eligible for bariatric surgery under the NHS.
* Diagnosed with impaired glucose regulation or type 2 diabetes, according to WHO 2011 criteria.
* Those with diabetes should be stable and well controlled with either diet or one oral hypoglycaemic agent.
* HbA1c ≤9.0% or 74.9 mmol/mol.

Exclusion criteria

* History of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer.
* Without access at home to a telephone or other factor likely to interfere with ability to participate reliably in the study.
* Pregnancy or breastfeeding.
* Smokers.
* Unable to maintain adequate contraception for the duration of the study and for one month afterwards.
* History of hypersensitivity to any of the components of the subcutaneous infusions.
* Donated blood during the preceding 3 months or intention to do so before the end of the study.
* Insulin treatment.
* Uncontrolled hypertension.
* Any other co-morbidity that would compromise the validity of the study or the safety of the participant such as heart failure, clinically apparent cardiovascular disease.
* Volunteers on anti-coagulants such as warfarin and factor Xa inhibitors will not undergo adipose tissue biopsy.
* Unable to give informed consent.
* Previous bariatric surgery.
* Unable to undergo fMRI due to:

  * Claustrophobia.
  * Pacemaker, metal implant, clips, implanted device, shrapnel or bullet, metal in eyes that precludes magnetic resonance imaging.
  * Significant structural abnormality on magnetic resonance brain scan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2013-10; Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Baseline - 4 weeks
  Weight loss as measured at baseline compared to 4 weeks after infusion or diet

SECONDARY OUTCOMES:
Glycaemia | Baseline - 4 weeks
  As assessed by change in fructosamine and HbA1c levels

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Bloom, FRS FRCP MD, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial CRF, Hammersmith Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available

REFERENCES:
- [Background] Alexiadou K, Cuenco J, Howard J, Wewer Albrechtsen NJ, Ilesanmi I, Kamocka A, Tharakan G, Behary P, Bech PR, Ahmed AR, Purkayastha S, Wheller R, Fleuret M, Holst JJ, Bloom SR, Khoo B, Tan TM. Proglucagon peptide secretion profiles in type 2 diabetes before and after bariatric surgery: 1-year prospective study. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e001076. doi: 10.1136/bmjdrc-2019-001076. PMID 32209584
- [Background] Ilesanmi I, Tharakan G, Alexiadou K, Behary P, Alessimii H, Bovill-Taylor C, Kenkre J, Choudhury S, Doyle C, Purkayastha S, Miras A, Tsironis C, Chahal H, Bloom SR, Oliver NS, Ahmed AR, Khoo B, Tan TM. Roux-en-Y Gastric Bypass Increases Glycemic Variability and Time in Hypoglycemia in Patients With Obesity and Prediabetes or Type 2 Diabetes: A Prospective Cohort Study. Diabetes Care. 2021 Feb;44(2):614-617. doi: 10.2337/dc20-1609. Epub 2020 Dec 17. PMID 33334806
- [Result] Behary P, Tharakan G, Alexiadou K, Johnson N, Wewer Albrechtsen NJ, Kenkre J, Cuenco J, Hope D, Anyiam O, Choudhury S, Alessimii H, Poddar A, Minnion J, Doyle C, Frost G, Le Roux C, Purkayastha S, Moorthy K, Dhillo W, Holst JJ, Ahmed AR, Prevost AT, Bloom SR, Tan TM. Combined GLP-1, Oxyntomodulin, and Peptide YY Improves Body Weight and Glycemia in Obesity and Prediabetes/Type 2 Diabetes: A Randomized, Single-Blinded, Placebo-Controlled Study. Diabetes Care. 2019 Aug;42(8):1446-1453. doi: 10.2337/dc19-0449. Epub 2019 Jun 8. PMID 31177183
- [Derived] Behary P, Alessimii H, Miras AD, Tharakan G, Alexiadou K, Aldhwayan MM, Purkayastha S, Moorthy K, Ahmed AR, Bloom SR, Tan TM. Tripeptide gut hormone infusion does not alter food preferences or sweet taste function in volunteers with obesity and prediabetes/diabetes but promotes restraint eating: A secondary analysis of a randomized single-blind placebo-controlled study. Diabetes Obes Metab. 2023 Jun;25(6):1731-1739. doi: 10.1111/dom.15028. Epub 2023 Mar 13. PMID 36811311
- [Derived] Kowalka AM, Alexiadou K, Cuenco J, Clarke RE, Minnion J, Williams EL, Bech P, Purkayastha S, Ahmed AR, Takats Z, Whitwell HJ, Romero MG, Bloom SR, Camuzeaux S, Lewis MR, Khoo B, Tan TM. The postprandial secretion of peptide YY1-36 and 3-36 in obesity is differentially increased after gastric bypass versus sleeve gastrectomy. Clin Endocrinol (Oxf). 2023 Sep;99(3):272-284. doi: 10.1111/cen.14846. Epub 2022 Nov 28. PMID 36345253
- [Derived] Jones B, Sands C, Alexiadou K, Minnion J, Tharakan G, Behary P, Ahmed AR, Purkayastha S, Lewis MR, Bloom S, Li JV, Tan TM. The Metabolomic Effects of Tripeptide Gut Hormone Infusion Compared to Roux-en-Y Gastric Bypass and Caloric Restriction. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e767-e782. doi: 10.1210/clinem/dgab608. PMID 34460933